CLINICAL TRIAL: NCT02416284
Title: Compliance to the Norwegian Food-Based Dietary Guidelines in Young Females
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oslo (Other)
Responsible Party: Principal Investigator, Rune Blomhoff, Professor, University of Oslo
Allocation: Not Applicable | Model: Single Group | Masking: Single
Other Study IDs: ERN4120_2012
Record Dates: First submitted 2015-04-03; First posted 2015-04-15 (Estimated); Last update posted 2015-04-15 (Estimated); Status verified 2015-04

CONDITIONS: Dietary Modification

STUDY DESIGN:
Who Masked: Participant

ARMS (1):
- NFBDG (Experimental): Multi-faceted, 2 week intervention to increase compliance to the NFBDG.
  Interventions: Other: NFBDG

INTERVENTIONS:
Other: NFBDG — Intervention consists of:
  Lecture presenting the NFBDG, Printed booklet containing the NFBDG, Suggested meal plan for a week, Recipes, Access to a restricted website with further information on the NFBDG, A Facebook-group where "Vegetable of the day" was presented with a suggested recipe, text-messages with encouragement to follow the guidelines, follow-up phone-calls, common exercise sessions, Free common meals (1 breakfast, 2 lunches, 1 dinner), Free foods (low-fat dairy products, a juice containing grapes, blueberries, chokeberries, and cherries and fruits)

SUMMARY:
The Norwegian Directorate of Health recently published the Norwegian food-based dietary guidelines (NFBDG) in 2011. The target for the NFBDG is the general population, and the main aims of these guidelines are to promote public health and prevent chronic degenerative diseases. Reaching the healthy population is crucial as only small proportion of the general population comply to the current public dietary advice in Norway. Thus, the objective of this study is to investigate whether a multi-faceted dietary intervention could increase compliance to the NFBDG and affect biomarkers of chronic degenerative diseases in a healthy population.

DETAILED DESCRIPTION:
The study was conducted as part of a master level course in Clinical Nutrition at the University of Oslo. Thus, the main objective of the study was to teach the master students about planning, conducting and analysing data from a clinical trial. The students themselves are subjects of the study, however the participation in the study was voluntary and did in no way affect the approval of the course.

Since the primary objective of the study was teaching, the study was confirmed by the "Regional Committees for Medical and Health Research Ethics" (REC) to be exempt from REC approval.

ELIGIBILITY:
Inclusion Criteria:

* female

Exclusion Criteria:

* serious chronic disease requiring medication
* pregnancy

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2012-09; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Biomarker of the intake of fruits and vegetables (caroteniods in plasma (uM) | 2 weeks
Biomarker of intake of fatty fish and low fat dairy products (fatty acids in red blood cells (fatty acid in % of FAME) | 2 weeks
  fatty acids in red blood cells (fatty acid in % of FAME)
Biomarker of the intake of fruits and vegetables (total antioxidant status in plasma (RU) | 2 weeks

SECONDARY OUTCOMES:
Lipids in plasma (HDL, LDL, total cholesterol) | 2 weeks
  HDL, LDL, total cholesterol
Blood glucose | 2 weeks
Blood pressure | 2 weeks
  Blood pressure (mmHg)
Weight (body weight in kg) | 2 weeks
  body weight in kg
Body composition (bioelectrocal impedance analysis (BIA) | 2 weeks
  bioelectrocal impedance analysis (BIA)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oslo, Oslo, Norway